CLINICAL TRIAL: NCT06819501
Title: Hyperbaric Oxygen Therapy for Peripheral Neuropathy Due to Paclitaxel Analogs
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Kun Wang, Professor, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2024-1015-04
Record Dates: First submitted 2025-01-21; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancers
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hyperbaric Oxygen group (Experimental): Administration of 100% oxygen at a pressure of 2.0ATA once daily for 60-90 minutes for a total of 30-40 times and administration of pressurised ice gloves 30 minutes before, during and 30 minutes after the administration of paclitaxel-based chemotherapeutic agents.
  Interventions: Device: hyperbaric oxygenation treatment; Behavioral: routine care
- Control group (Active Comparator): Administration of pressurised ice gloves 30 minutes before, during, and 30 minutes after administering paclitaxel chemotherapy drugs.
  Interventions: Behavioral: routine care

INTERVENTIONS:
Device: hyperbaric oxygenation treatment — Administration of 100% oxygen at a pressure of 2.0ATA once daily for 60-90 minutes for a total of 30-40 times.
  Arms: Hyperbaric Oxygen group
Behavioral: routine care — Administration of pressurised ice gloves 30 minutes before, during, and 30 minutes after administering paclitaxel chemotherapy drugs.

SUMMARY:
The goal of this study was to explore the safety and efficacy of hyperbaric oxygen in the treatment of peripheral neuropathy due to paclitaxel analogues

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly diagnosed breast cancer by pathology
2. Age 18-60 years
3. ECOG 0-2
4. CIPN patients with NCI-CTCAE grade 1 or higher after treatment with paclitaxel-based drugs

Exclusion Criteria:

1. Patients with contraindications to hyperbaric oxygen i. Untreated pneumothorax. ii. concomitant administration of disulfiram. iii. concomitant administration of antineoplastic drugs such as bleomycin, cisplatin, adriamycin. iv. premature and/or low body mass newborns.

   iv. Premature and/or low body mass neonates.
2. Other cancers

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 226 (Estimated)
Dates: Start 2025-02-05 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Difference in change in CIPN score due to paclitaxel analogues compared to baseline | Baseline, 2 week, 4 week, 6 week, 8 week
  Difference in change in CIPN score due to paclitaxel analogues compared to baseline

SECONDARY OUTCOMES:
NPS degree | Baseline, 2 week, 4 week, 6 week, 8 week
EORTC QLQ - CIPN20 | Baseline, 2 week, 4 week, 6 week, 8 week
ENS score | Baseline, 2 week, 4 week, 6 week, 8 week
neuromyography | Baseline, 8 week
life quality | Baseline, 2 week, 4 week, 6 week, 8 week
  FACT-B Quality of Life Score
insomnia score | Baseline, 2 week, 4 week, 6 week, 8 week
  Insomnia Severity Index (ISI)
depression score | Baseline, 2 week, 4 week, 6 week, 8 week
  Hospital Anxiety and Depression Scale (HADS)
Exhaustion score | Baseline, 2 week, 4 week, 6 week, 8 week
  Brief Fatigue Inventory (BFI)
Side effects of hyperbaric oxygen therapy | during the hyperbaric oxygen therapy (up to 2 months)

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China